CLINICAL TRIAL: NCT01194167
Title: A Phase II Study of Eltrombopag in Platelet Refractory Thrombocytopenia
Brief Title: Study of Eltrombopag in Platelet Refractory Thrombocytopenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to identify eligible patients
Sponsor: University of Cincinnati (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCC-H1
Record Dates: First submitted 2010-08-25; First posted 2010-09-02 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2012-01

CONDITIONS: Thrombocytopenia
Keywords: Platelet refractory thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — eltrombopag

ARMS (1):
- Eltrombopag (Experimental): Eltrombopag 75 mg per day. Possible escalation to 150 mg per day after day 15 lab results. Possible escalation to 300 mg per day after day 29 lab results.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — 75 mg per day with possible dose escalation to 150 mg per day and 300 mg per day

SUMMARY:
This phase II trial is studying the effects of the drug eltrombopag has on thrombocytopenia (low platelet count). Eltrombopag is approved by the FDA for the treatment of thrombocytopenia (low platelet count) in adults who have had an insufficient response to medications such as corticosteroids and immunoglobulins. Eltrombopag is not approved by the FDA (Food and Drug Administration) for the treatment of thrombocytopenia refractory to platelet transfusion and so for this study is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory diagnosis of platelet refractoriness
* Diagnosis of platelet dependence
* Adequate liver and renal laboratory screening tests

Exclusion Criteria:

* Patients with thrombocytopenia that are responsive to platelet therapy
* Patients actively receiving intravenous immunoglobulin, plasmapheresis or cytotoxic medications for thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determine the likelihood of eltrombopag allowing platelet transfusion independence in patients with platelet refractoriness at doses of 75 mg, 150 mg, and 300 mg per day | 3 years average

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Carey, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States